CLINICAL TRIAL: NCT07267182
Title: Comparative Efficacy of Gabapentin and Diclofenac Sodium for Post-Operative Pain Relief in Patients Undergoing Major Abdominal Surgeries
Brief Title: Gabapentin and Diclofenac Sodium Comparison for Post-Operative Pain Relief
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Muhammad Aamir Latif (Other)
Responsible Party: Sponsor-Investigator, Muhammad Aamir Latif, Research Consultant, RESnTEC, Institute of Research
Organization: RESnTEC, Institute of Research (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DR-SAIMA-QAMC
Record Dates: First submitted 2025-11-24; First posted 2025-12-05 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Gabapentin; Diclofenac

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gabapentin group (Experimental): Patients received a single oral dose of gabapentin 600 mg one hour before surgery.
  Interventions: Drug: Gabapentin 600mg
- Diclofenac group (Experimental): Patients were given a single oral dose of diclofenac sodium 100 mg one hour before surgery.
  Interventions: Drug: Diclofenac Sodium 100 MG

INTERVENTIONS:
Drug: Gabapentin 600mg — Patients received a single oral dose of gabapentin 600 mg one hour before surgery.
  Arms: Gabapentin group
Drug: Diclofenac Sodium 100 MG — Patients were given a single oral dose of diclofenac sodium 100 mg one hour before surgery.
  Arms: Diclofenac group

SUMMARY:
Little is known about comparative efficacy of gabapentin and diclofenac sodium in managing post-operative pain. Therefore, this study was planned to compare the efficacy of gabapentin, and diclofenac sodium for post-operative pain relief in patients undergoing major abdominal surgeries.

DETAILED DESCRIPTION:
Non-steroidal anti-inflammatory drugs, opioid analgesics, and local and regional anesthesia have been used as preventive interventions, but their role in postoperative pain management remains inconclusive. Gabapentin is a relatively new drug for postoperative pain management whose side effects are well tolerated. If the findings of this study produce similar observations, it would add to the already scarce data and help patients undergoing major abdominal surgeries in the local settings in relieving postoperative pain effectively.

ELIGIBILITY:
Inclusion Criteria:

* Any gender
* Aged 18-60 years
* Undergoing elective major abdominal surgery under general anesthesia
* With physical status I or II
* Who were able to comprehend and use the Visual Analogue Scale (VAS) for pain assessment

Exclusion Criteria:

* With a known allergy or contraindication to gabapentin, or diclofenac sodium
* A history of peptic ulcer disease
* A history of gastrointestinal bleeding
* Hepatic or renal dysfunction
* Pregnancy or lactation
* With neurological or psychiatric disorders affecting pain perception
* Received opioids, anticonvulsants, antidepressants, or nonsteroidal anti-inflammatory drugs (NSAIDs) within 24 hours before surgery
* With uncontrolled hypertension, ischemic heart disease, or diabetes mellitus
* Those who experienced intraoperative complications necessitating a change in anesthetic plan or postoperative mechanical ventilation

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 240 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-02-28 (Actual)

PRIMARY OUTCOMES:
Pain reduction | 12 hours
  Patients were considered to have effective pain relief ("Yes") if their VAS score remained ≤3 throughout the monitoring period without requiring rescue analgesia.

CONTACTS AND LOCATIONS:
Overall Officials: Saima Noreen, Principal Investigator — Quid-e-Azam Medical College, Bahawalpur; Ambreen Khan, Principal Investigator — Quid-e-Azam Medical College, Bahawalpur; Qazi Anees, Principal Investigator — Quid-e-Azam Medical College, Bahawalpur
Locations (1):
- Bahawal Victoria Hospital, Bahawalpur, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No
Data can be shared on a reasonable request.